CLINICAL TRIAL: NCT06968871
Title: Effects of the Ameliorated Pap Test on Cervical Cancer Screening Participation: a Multicenter Randomized Controlled Trial
Brief Title: Ameliorated Pap Tests and Cervical Cancer Screening Participation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); National Taiwan University (Other); National Taiwan University Hospital Beihu Branch (Other); National Taiwan University Hospital, Yun-Lin Branch (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 202502041RINE
Record Dates: First submitted 2025-04-27; First posted 2025-05-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Screening; Cervical Cancer Screening Methods
Keywords: Cancer screening participation; Cervical cancer; Multicenter; Multidisciplinary; Pain; Pap smear; Peak-end concept; Preventive medicine; Randomized controlled trial
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Cytopathologists who analyze the specimens are blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Pap test (No Intervention)
- Modified Pap test (Experimental)
  Interventions: Procedure: Modified Pap test

INTERVENTIONS:
Procedure: Modified Pap test — For the intervention group receiving the modified Pap test, instead of immediately removing the speculum just after rotating back the speculum, an operator still fixes the speculum in the vagina for 15 seconds.
  Arms: Modified Pap test

SUMMARY:
The Pap test plays a crucial role in the early detection of cervical cancer. A pilot single-center randomized controlled trial applied the peak-end concept and added a non-painful step at the end of Pap smear screening, aimed to reduce recalled pain. However, there is still no multicenter study investigating the effect of the modified Pap test on cervical cancer screening participation.

The present project is the first multicenter randomized controlled trial to expand the current scope of the peak-end theory into Pap tests and cervical cancer screening participation by adding a non-painful step at the end of Pap smear screening. Our multidisciplinary team (NTUH Pap Study Group) aims to provide innovative, feasible, and low-cost strategies for cervical cancer screening participation.

DETAILED DESCRIPTION:
Participants: This project expects to include women just before they undergo Pap smear screening at the NTUH Healthcare System in 2026. We include eligible women aged 25 or above who have not yet undergone Pap tests in 2026. Excluded are those who have ongoing menstruation and those who are pregnant or incapable of understanding the numeric pain scales. Women who have any active cancer at study entry (defined as cancer diagnosed or treated within the previous 6 months, recurrent, regionally advanced or metastatic cancer), previous hysterectomy, previous pelvic surgery or radiotherapy, active vaginal or uterus infection, and analgesic use within 24 hours are excluded due to potential interference with pain intensity. The study protocol was approved by the NTUH Research Ethics Committee. During the recruitment process, every eligible participant is fully informed of this trial's aim, design, and content, except for the intervention details. All participants should provide written informed consent. This study is conducted according to the Declaration of Helsinki and is registered at ClinicalTrials.gov.

Sample size estimation: The investigators estimate to recruit at least 248 participants (180 at the NTUH, 68 at the NTUH Hsin-Chu, Bei-Hu, Yunlin, and Cancer Center branches), 50% (124) of whom are randomized to the intervention group, to reach 90% power for the detection of an increase in 3-year cervical cancer screening participation from 30% to 50% at the 5% level of significance.

Randomization and blinding: Eligible participants are randomly assigned to either the group receiving the traditional Pap test or the modified Pap test. Computer-generated random numbers are employed for simple randomization with a 1:1 allocation ratio. All participants are kept unaware of any information about group allocation throughout the study period. The operators performing the procedure are not informed by the assistants whether to intervene until a specimen is prepared for cervical cytology. The delayed disclosure of the group allocation until this step ensures that the operators standardize the insertion and opening phases of the Pap test. Cytopathologists who analyze the specimens are blinded to the study.

The modified and traditional Pap tests: All operators experienced in techniques for performing a Pap test should attend workshops for a standard operating procedure. The operators include family physicians and gynecologists. A well-trained research assistant is also responsible for ensuring standardization of procedures to eliminate interoperator variability. During the Pap test, there is a privacy curtain separating participants from the operators. An operator separates the labia with hand and then gently inserts the saline-lubricated speculum sideways. The speculum is rotated 90 degrees and opened to achieve an optimal view of the cervix. Then an operator fixes the speculum to obtain the cell samples by brushes. The above-standardized procedures are the same between the two groups. After preparing a specimen for conventional cytology, an operator loosens the locking nut of the speculum, partially closes the blade, rotates the speculum 90 degrees back to its original insertion orientation, and then removes the speculum in the control group receiving the traditional Pap test. For the intervention group receiving the modified Pap test, instead of immediately removing the speculum just after rotating back the speculum, an operator still fixes the speculum in the vagina for 15 seconds. Participants receiving the modified Pap test do not realize what is going on during the 15-second step because they are behind the privacy curtain. Procedurally, the subsequent addition of a non-painful step after specimen collection does not affect specimen quality.

Interview, Anthropometric Indices, and Anxiety scores: The investigators review the medical records after getting informed consent. In addition to pain evaluations, this project collects information about tobacco use, alcohol consumption, socioeconomic status, marital status, parity, sexually active status, menopause, predicted pain of Pap smears, psychological stress, anxiety score, analgesic use, current medications, and medical history through standardized personal interviews. Body height and weight are measured using a standard stadiometer, and body mass index is calculated. Blood pressure is measured with an electronic sphygmomanometer while the patient is seated after resting for at least five minutes. Psychological stress is assessed using the Brief Symptom Rating Scale -5 (BSRS-5). The BSRS-5 includes items of anxiety, depression, hostility, interpersonal sensitivity, and insomnia measured by a 5-point Likert-type scale of 0-4. Normal, slight, and great mental stress is defined by the sum of BSRS-5 scores ≤ 5, 6-9, and ≥10, respectively. The anxiety score is obtained using the Generalized Anxiety Disorder 7-item (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21 (0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety). Based on a meta-analysis, some experts have recommended considering using a cut-off of 8 to optimize sensitivity without compromising specificity.

Statistical analyses: For the descriptive analyses, values are presented as either numbers (percentages) or mean ± standard deviations. For the univariate analyses, categorical data are compared by the χ2 or Fisher's exact tests. Continuous data are compared using the independent T test. To compare screening uptake between trial groups, the investigators apply an ITT principle, such that outcomes are analyzed according to the trial groups assigned, regardless of whether the participants comply with the intervention components of each trial group. Logistic regression analyses are utilized to estimate the association of the intervention with the probability of 3-year and 1-year uptake of cervical cancer screening. The investigators use the five-region hypothesis test based on odds ratios to test the significant indistinguishability of real-time pain between the two groups for confirming the success of randomization and blinding. The effect sizes of five-minute recalled pain on a 1-5 numeric scale and a 0-10 VAS between the two groups are calculated using Glass's delta. Linear regression analyses are used to estimate the effect of the intervention on scores of 5-minute and 3-month recalled pains. Prespecified subgroup analyses using both linear and logistic regression analyses will be performed and summarized visually using forest plots. Major subgroups of interest include women who are never screened (never underwent Pap tests) and women who are under-screened (have not undergone Pap tests in the past 3 years). Statistical significance levels are determined by two-tailed tests (P < 0.05). The statistical analyses are performed with SAS software version 9.4 (SAS Institute Inc., Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 or above

Exclusion Criteria:

* Ongoing menstruation
* Pregnancy
* Incapability of understanding the numeric pain scales
* Any active cancer at study entry (defined as cancer diagnosed or treated within the previous 6 months, recurrent, regionally advanced or metastatic cancer)
* Previous hysterectomy, pelvic surgery, or radiotherapy
* Active vaginal or uterus infection
* Analgesic use within 24 hours

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year cervical cancer screening participation | 3 years
  Defined as attending a Pap test at any clinic before the end of the 3rd subsequent year following study entry

SECONDARY OUTCOMES:
1-year cervical cancer screening participation | 1 year
  Defined as attending a Pap test at any clinic before the end of the next year following study entry
5-minute recalled pain intensity on a 1-5 numeric scale and a 0-10 visual analog scale | 5 minutes after receiving the Pap smear test
  Recalled pain intensity at 5 minutes after the Pap smear test with evaluation by a 1-5 numeric scale and a 0-10 visual analog scale.
3-month recalled pain intensity on a 1-5 numeric scale and a 0-10 visual analog scale | 3 months after receiving the Pap smear test
  Recalled pain intensity at 3 months after the Pap smear test with evaluation by a 1-5 numeric scale and a 0-10 visual analog scale. To minimize potential propaganda for cervical cancer screening participation, the investigators choose the 3-month interval rather than 6-month or 1-year intervals for long-term pain recollection after Pap tests.
Real time pain during the Pap test using a 1-5 numeric scale | Every five seconds throughout the Pap test, up to completion of Pap test
  The participants will evaluate and record their pain every five seconds throughout the test with an application on a 1 to 5 numeric scale. The average pain, the maximal pain, and real-time pain at the beginning, first quarter, second quarter, third quarter, and the end of the regular course are compared between the two groups. The investigators will compare the average pain of each group's first and second half of the course's course. For participants receiving the modified Pap test, the investigators further compare the average pain, the maximal pain, and the last recorded real-time pain of the 15-second step with that of the regular course.

OTHER OUTCOMES:
Patient-reported feedback at the end of the study | At the fourth follow-up year in participants who do not undergo the 3-year cervical cancer screening; or between 1 and 12 months after the latest Pap test in participants who undergo the 3-year cervical cancer screening
  Patient-reported feedback at the health-service level drives revolutions and innovations. At the end of the study period (after the end of the third follow-up year in participants who do not undergo the 3-year cervical cancer screening after the study entry; or at least one month after the latest Pap test in participants who undergo the 3-year cervical cancer screening after the study entry), all participants will be asked to provide open-ended feedback for future qualitative research on Pap smear screening (detailed in subsequent research proposals). For instance, "Can you tell me more about your thoughts on Pap tests you have undergone these years?" or "What is your opinion on the future of Pap tests?".

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsieh Chiang, MD, MPH, PhD, Study Chair — National Taiwan University Hospital & College of Medicine
Locations (5):
- Taiwan (5):
  - National Taiwan University Hospital Yunlin Branch, Douliu
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei
  - National Taiwan University Hospital Beihu Branch, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jhuang JR, Lee WC, Chan CC. A randomized, double-blind water taste test to evaluate the equivalence of taste between tap water and filtered water in the Taipei metropolis. Sci Rep. 2020 Aug 7;10(1):13387. doi: 10.1038/s41598-020-70272-y. PMID 32770131
- [Background] Shih HY, Lee WC. A Five-Region Hypothesis Test for Exposure-Disease Associations. Sci Rep. 2017 Jul 11;7(1):5131. doi: 10.1038/s41598-017-05301-4. PMID 28698548
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Chen HC, Wu CH, Lee YJ, Liao SC, Lee MB. Validity of the five-item Brief Symptom Rating Scale among subjects admitted for general health screening. J Formos Med Assoc. 2005 Nov;104(11):824-9. PMID 16496062
- [Background] Chen CJ, Hong MK, Ding DC. Effective reduction in inadequate Pap smears by using a saline-lubricated speculum and two glass slides. Taiwan J Obstet Gynecol. 2020 Nov;59(6):906-909. doi: 10.1016/j.tjog.2020.09.018. PMID 33218410
- [Background] Sandkuhler J, Lee J. How to erase memory traces of pain and fear. Trends Neurosci. 2013 Jun;36(6):343-52. doi: 10.1016/j.tins.2013.03.004. Epub 2013 Apr 18. PMID 23602194
- [Background] Yen HK, Cheng SY, Chiu KN, Huang CC, Yu JY, Chiang CH; NTUH Pap Study Group. Adding a nonpainful end to reduce pain recollection of Pap smear screening: a randomized controlled trial. Pain. 2023 Aug 1;164(8):1709-1717. doi: 10.1097/j.pain.0000000000002897. Epub 2023 Apr 12. PMID 37043729
- [Background] Hsu CF, Propp L, Panetta L, Martin S, Dentakos S, Toplak ME, Eastwood JD. Mental effort and discomfort: Testing the peak-end effect during a cognitively demanding task. PLoS One. 2018 Feb 12;13(2):e0191479. doi: 10.1371/journal.pone.0191479. eCollection 2018. PMID 29432429
- [Background] Muller UWD, Witteman CLM, Spijker J, Alpers GW. All's Bad That Ends Bad: There Is a Peak-End Memory Bias in Anxiety. Front Psychol. 2019 Jun 12;10:1272. doi: 10.3389/fpsyg.2019.01272. eCollection 2019. PMID 31249540
- [Background] Schneider S, Stone AA, Schwartz JE, Broderick JE. Peak and end effects in patients' daily recall of pain and fatigue: a within-subjects analysis. J Pain. 2011 Feb;12(2):228-35. doi: 10.1016/j.jpain.2010.07.001. PMID 20817615
- [Background] Arney J, Hinojosa-Lindsey M, Street RL Jr, Hou J, El-Serag HB, Naik AD. Patient experiences with surveillance endoscopy: a qualitative study. Dig Dis Sci. 2014 Jul;59(7):1378-85. doi: 10.1007/s10620-014-3035-4. Epub 2014 Feb 6. PMID 24500449
- [Background] Redelmeier DA, Katz J, Kahneman D. Memories of colonoscopy: a randomized trial. Pain. 2003 Jul;104(1-2):187-94. doi: 10.1016/s0304-3959(03)00003-4. PMID 12855328
- [Background] Redelmeier DA, Kahneman D. Patients' memories of painful medical treatments: real-time and retrospective evaluations of two minimally invasive procedures. Pain. 1996 Jul;66(1):3-8. doi: 10.1016/0304-3959(96)02994-6. PMID 8857625
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Lin SN, Taylor J, Alperstein S, Hoda R, Holcomb K. Does speculum lubricant affect liquid-based Papanicolaou test adequacy? Cancer Cytopathol. 2014 Mar;122(3):221-6. doi: 10.1002/cncy.21369. Epub 2013 Nov 19. PMID 24254917
- [Background] Uygur D, Guler T, Yayci E, Atacag T, Comunoglu C, Kuzey GM. Association of speculum lubrication with pain and Papanicolaou test accuracy. J Am Board Fam Med. 2012 Nov-Dec;25(6):798-804. doi: 10.3122/jabfm.2012.06.120021. PMID 23136318
- [Background] Keskin AE, Onaran Y, Duvan IC, Simavli S, Kafali H. Topical anesthetic (lidocaine-prilocaine) cream application before speculum examination in postmenopausal women. J Minim Invasive Gynecol. 2012 May-Jun;19(3):350-5. doi: 10.1016/j.jmig.2012.01.005. Epub 2012 Mar 13. PMID 22417905
- [Background] Simavli S, Kaygusuz I, Kinay T, Cukur S. The role of gel application in decreasing pain during speculum examination and its effects on papanicolaou smear results. Arch Gynecol Obstet. 2014 Apr;289(4):809-15. doi: 10.1007/s00404-013-3047-x. Epub 2013 Oct 12. PMID 24121692
- [Background] Leung SS, Leung I. Cervical cancer screening: knowledge, health perception and attendance rate among Hong Kong Chinese women. Int J Womens Health. 2010 Aug 9;2:221-8. doi: 10.2147/ijwh.s10724. PMID 21072314
- [Background] Song W, Li H, Sun F, Guo T, Jiang S, Wang X. Pain Avoidance and Its Relation to Neural Response to Punishment Characterizes Suicide Attempters with Major Depression Disorder. Psychiatry Res. 2020 Dec;294:113507. doi: 10.1016/j.psychres.2020.113507. Epub 2020 Oct 13. PMID 33075650
- [Background] Claes N, Crombez G, Vlaeyen JWS. Pain-avoidance versus reward-seeking: an experimental investigation. Pain. 2015 Aug;156(8):1449-1457. doi: 10.1097/j.pain.0000000000000116. PMID 25775360
- [Background] Gauss JW, Mabiso A, Williams KP. Pap screening goals and perceptions of pain among black, Latina, and Arab women: steps toward breaking down psychological barriers. J Cancer Educ. 2013 Jun;28(2):367-74. doi: 10.1007/s13187-012-0441-1. PMID 23288606
- [Background] Hoyo C, Yarnall KS, Skinner CS, Moorman PG, Sellers D, Reid L. Pain predicts non-adherence to pap smear screening among middle-aged African American women. Prev Med. 2005 Aug;41(2):439-45. doi: 10.1016/j.ypmed.2004.11.021. PMID 15917039
- [Background] Masson H. Cervical pap smears and pandemics: The effect of COVID-19 on screening uptake & opportunities to improve. Womens Health (Lond). 2021 Jan-Dec;17:17455065211017070. doi: 10.1177/17455065211017070. PMID 34032158
- [Background] Holroyd E, Twinn S, Adab P. Socio-cultural influences on Chinese women's attendance for cervical screening. J Adv Nurs. 2004 Apr;46(1):42-52. doi: 10.1111/j.1365-2648.2003.02964.x. PMID 15030441
- [Background] Kaneko N. Factors associated with cervical cancer screening among young unmarried Japanese women: results from an internet-based survey. BMC Womens Health. 2018 Jul 31;18(1):132. doi: 10.1186/s12905-018-0623-z. PMID 30064505
- [Background] Friedman AM, Hemler JR, Rossetti E, Clemow LP, Ferrante JM. Obese women's barriers to mammography and pap smear: the possible role of personality. Obesity (Silver Spring). 2012 Aug;20(8):1611-7. doi: 10.1038/oby.2012.50. Epub 2012 Feb 28. PMID 22370590
- [Background] Chou HH, Huang HJ, Cheng HH, Chang CJ, Yang LY, Huang CC, Chang WY, Hsueh S, Chao A, Wang CJ, Tang YH, Lin CT, Qiu JT, Chen MY, Chen CY, Huang KG, Tsai TC, Chang TC, Lai CH. Self-sampling HPV test in women not undergoing Pap smear for more than 5 years and factors associated with under-screening in Taiwan. J Formos Med Assoc. 2016 Dec;115(12):1089-1096. doi: 10.1016/j.jfma.2015.10.014. Epub 2015 Dec 23. PMID 26723863
- [Background] Yang CM, Sung FC, Hsue CS, Muo CH, Wang SW, Shieh SH. Comparisons of Papanicolaou Utilization and Cervical Cancer Detection between Rural and Urban Women in Taiwan. Int J Environ Res Public Health. 2020 Dec 28;18(1):149. doi: 10.3390/ijerph18010149. PMID 33379209
- [Background] Sirovich BE, Welch HG. The frequency of Pap smear screening in the United States. J Gen Intern Med. 2004 Mar;19(3):243-50. doi: 10.1111/j.1525-1497.2004.21107.x. PMID 15009779
- [Background] Dugue PA, Lynge E, Rebolj M. Mortality of non-participants in cervical screening: Register-based cohort study. Int J Cancer. 2014 Jun 1;134(11):2674-82. doi: 10.1002/ijc.28586. Epub 2013 Nov 29. PMID 24288241
- [Background] Andrae B, Andersson TM, Lambert PC, Kemetli L, Silfverdal L, Strander B, Ryd W, Dillner J, Tornberg S, Sparen P. Screening and cervical cancer cure: population based cohort study. BMJ. 2012 Mar 1;344:e900. doi: 10.1136/bmj.e900. PMID 22381677